CLINICAL TRIAL: NCT06400420
Title: The Effect of Classical Futsal Training Program on Physical Fitness Level of University Amateur Futsal Players
Brief Title: The Effect of Futsal Training on Physical Fitness in Amateur Futsal Players
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Bilal Deniz Aydos, Bilal Deniz Aydos, Istanbul Medipol University Hospital
Other Study IDs: E-10840098-604.01.01-1310
Record Dates: First submitted 2024-02-25; First posted 2024-05-06 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Futsal; Physical Fitness
Keywords: Futsal; Physical fitness; risk analysis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exercise — classic futsal training program

SUMMARY:
The goal of this observational study is to examine the effects of classical futsal training on physical fitness in amateur futsal players. The main question[s] it aims to answer are:

• Does classical futsal training have any effect on the physical fitness level of futsal players? Participants will be taken to the classical futsal training program for 8 weeks. Before and after 8 weeks, players will be evaluated for their physical fitness.

DETAILED DESCRIPTION:
The study was planned to be carried out as a non-randomized clinical study with 30 athletes in the university futsal team.

All athletes will be evaluated at the beginning of the training and will continue their classical futsal training for 8 weeks.

The program to be applied in addition to routine training 2 times a week;

* It will begin with a 10-minute standard futsal workout warm-up. warm-up program; It will consist of light aerobic exercises and dynamic stretching of large muscle groups.
* After the warm-up period, all groups will participate in the standard 45-minute futsal training.
* Finally, the training will end with 5 minutes of cool-down exercises (dynamic stretching).

The first evaluation will be made 2 days before the athletes' routine training, and the next evaluations will be made at least 2 days after the last training.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-25
* Playing in Istanbul Medipol University futsal team
* 2 days a week, 2 hours training for futsal or 1 game a week and 2 hours a week, 2 days a week

Exclusion Criteria:

* History of lower extremity injury or surgery within 6 months prior to the test
* Injury three months before the study,
* Failure to heal or complete rehabilitation of previous injury,
* Physical or mental conditions that prevent them from participating in technical and tactical futsal training and/or experimental training programs
* Two or more missed training sessions

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Male athletes between the ages of 18-25, who are in the Istanbul Medipol University Futsal team, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in balance after 8-week training program | 8 Week
  Y Balance Test
Change in muscle strenght after 8-week training program | 8 week
  Myometer Measurement
Change in anaerobic capacity after 8-week training program | 8 week
  Running Based Anaerobic Sprint Test
Change in flexibility after 8-week training program | 8 week
  Sit and Reach Test
Change in stability after 8-week training program | 8 week
  Closed kinetic chain lower extremity stability test

CONTACTS AND LOCATIONS:
Locations (1):
- Bİlal Deniz Aydos, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided